CLINICAL TRIAL: NCT07250568
Title: Effects of Exercise, Posture Education, and Standing Advice on Pain, Lumbar Posture, Core Stability, Flexibility, Fatigue, Endurance, Ergonomics, Stress, and Quality of Life in Office Workers With Low Back Pain: A Three-Arm RCT
Brief Title: Office Program Effects on Pain, Posture, Muscle Physiology, Stress, Ergonomics, and Quality of Life in LBP Workers
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Suci Wahyu Ismiyasa (Other)
Collaborators: Pembangunan Nasional Veteran Jakarta University (Other)
Responsible Party: Sponsor-Investigator, Suci Wahyu Ismiyasa, Supervisor: Zarina Zahari, PhD, University Teknologi MARA; Principal Investigator: Suci Wahyu Ismiyasa, M.Erg, Universiti Teknologi Mara
Organization: Universiti Teknologi Mara (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UTMara-OWP-LBP2025
Record Dates: First submitted 2025-11-16; First posted 2025-11-26 (Actual); Last update posted 2025-11-26 (Actual); Status verified 2025-11

CONDITIONS: Low Back Pain
Keywords: Low back pain; Office Workers; Ergonomics; Exercise Intervention; Posture Education
MeSH Terms: conditions — Low Back Pain | interventions — Exercise; Educational Status; Counseling

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned into three parallel intervention groups that differ in the components of the office worker's program they receive. The three groups will run concurrently throughout the study period. Exercise group will receive a combined intervention consisting of an exercise program, posture education, and standing advice. Education group will receive posture education and a standing advice. Control Group will receive only the standing advice as a minimal intervention control. Each participant remains in their assigned group for the duration of the study, and outcomes will be compared across groups to evaluate the relative effectiveness of each intervention combination.
Masking Description: No masking was performed. The study is open-label, and neither participants nor investigators were blinded to group assignment due to the nature of the intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Exercise Group (Experimental): Participants in this arm will receive a structured exercise program supervised by a physiotherapist, combined with posture education using an illustrated poster and regular standing advice. The exercise program consists of progressive abdominal and lumbar strengthening exercises performed 3 times per week for 12 weeks, with each session lasting approximately 20 minutes.
  Interventions: Behavioral: Exercise; Behavioral: Education; Behavioral: Advice
- Education Group (Active Comparator): Participants in this arm will receive posture education supported by an illustrated poster and regular standing advice. No exercise program will be provided to this group.
  Interventions: Behavioral: Education; Behavioral: Advice
- Control Group (Active Comparator): Participants in this arm will receive standing advice only, without exercise intervention or posture education materials.
  Interventions: Behavioral: Advice

INTERVENTIONS:
Behavioral: Exercise — Exercise Program: A structured physiotherapist-supervised exercise program designed to improve core stability, lumbar strength, flexibility, and endurance. The program includes progressive abdominal and lumbar muscle strengthening exercises performed three times per week for 12 weeks, with each session lasting approximately 20 minutes. Exercises gradually increase in intensity based on participant tolerance and progression criteria.
  Arms: Exercise Group
Behavioral: Education — An educational ergonomic intervention delivered using an illustrated posture guidance poster. Participants receive instruction on proper sitting posture, workstation alignment, neutral spine position, and strategies to reduce lumbar strain during daily office activities. Education is delivered at baseline with follow-up reminders throughout the 12-week study period.
  Other Names: Poster Education
  Arms: Education Group; Exercise Group
Behavioral: Advice — A behavioral intervention in which participants are advised to take regular standing breaks to reduce prolonged sitting. Participants are instructed to stand for short intervals periodically during working hours, supported by scheduled reminders. No exercise or posture education materials are included in this intervention.

SUMMARY:
This interventional study aims to evaluate the effectiveness of an office worker's program in reducing low back pain and improving physical and psychosocial outcomes among office employees. The primary objective is to determine the effects of the intervention on pain, lumbar posture, muscle physiology (including core stability, flexibility, fatigue, and endurance), ergonomics, stress levels, and quality of life across different intervention groups.

Participants will be assigned to one of three groups:

Group 1: Exercise program, posture education, and standing advice Group 2: Posture education and standing advice Group 3: standing advice only The study will compare outcomes between groups to identify which combination of interventions provides the greatest benefits for office workers with a tendency to experience low back pain.

DETAILED DESCRIPTION:
Research question: Is there any effect of office worker's program on pain intensity, lumbar posture, muscle physiology, ergonomics, stress and quality of life among office workers with low back pain? Research objective: To determine the effect of office worker's program on pain intensity, lumbar posture, muscle physiology, ergonomics, stress and quality of life Research hypothesis: There is significance different on pain intensity, lumbar posture, muscle physiology, ergonomics, stress and quality of life

ELIGIBILITY:
Inclusion Criteria:

1. Identified LBP
2. Age between 18 - 60 years old
3. In the office, working in front computer/laptop minimum along 4 hours per day
4. Able to ambulate independently with or without walking aids
5. Controlled comorbidity e.g. DM, HPT, managed asthma and controlled thyroid conditions

Exclusion Criteria:

1. Recumbent
2. Cancer, spinal fracture, neurological disorder (stroke, PBI and soon)
3. Participation in a current fitness program designed to prevent LBP recurrence
4. Spinal operation within the last six months
5. Pregnant
6. Medication (steroid therapy, non-steroidal anti-inflammatory drugs (NSAIDs), opioids, muscle relaxants, antidepressants or anxiolytics)
7. Insufficient to finish outcome measurements and exercise program
8. Participants who do not attend 3 consecutive weeks or 8 consecutive times

Ages: 18 Years to 58 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2026-03-23 (Estimated); Primary Completion 2026-06-17 (Estimated); Study Completion 2026-08-01 (Estimated)

PRIMARY OUTCOMES:
Numeric Rating Scale for pain | Baseline and Week 12
  Pain intensity will be assessed using the Numeric Rating Scale (NRS), an 11-point scale from 0 (no pain) to 10 (worst possible pain). Participants will rate their average low back pain at baseline and after the 12-week intervention. Changes in NRS scores will be compared across groups.

SECONDARY OUTCOMES:
Flexible curve to measure Lumbar posture | Baseline and Week 12
  Lumbar posture will be assessed using the Flexible Curve method, which measures lumbar curvature by molding a flexible ruler along the participant's lumbar spine. Measurements will be taken in the prone position to assess lumbar extension and in the sitting position to assess lumbar flexion. The molded curve will then be traced onto paper to calculate the lumbar lordosis angle and curvature index. Changes in lumbar curvature values will be compared between groups to determine the effects of the interventions on spinal alignment. The unit of measurement will be degrees.
Sphygmomanometer Pressure Test to measure Core Stability | Baseline and Week 12
  Core stability will be assessed using a sphygmomanometer pressure biofeedback test. Participants will be positioned sitting, with the cuff placed behind the lumbar region and inflated to a baseline pressure of 40 mmHg. Changes in pressure during controlled abdominal drawing-in maneuvers will be recorded. Smaller pressure deviations indicate better core muscle activation and stability. Core stability scores will be compared between groups to evaluate the effectiveness of each intervention. The unit of measurement will be millimeters of mercury (mmHg).
Short Form-36 (SF-36) to measure quality of life | Baseline and Week 12
  Quality of life will be assessed using the Short Form-36 (SF-36) questionnaire, which measures eight health domains: physical functioning, role limitations due to physical health, bodily pain, general health, vitality, social functioning, role limitations due to emotional problems, and mental health. Each domain is scored from 0 to 100, with higher scores indicating better health status. Changes in SF-36 scores will be compared between groups to determine the impact of the interventions on overall quality of life.
Perceived Stress Scale (PSS) to measure stress | Baseline and Week 12
  Stress levels will be assessed using the Perceived Stress Scale (PSS), a validated self-report questionnaire that measures the degree to which situations in a participant's life are appraised as stressful. Participants complete the 10-item PSS, with each item scored on a 0-4 scale. Higher total scores indicate higher perceived stress. Changes in PSS scores will be compared between the three study groups to evaluate the effect of the interventions on stress reduction.
Rapid Office Strain Assessment (ROSA) to measure ergonomics | Baseline and Week 12
  Ergonomic risk will be evaluated using the Rapid Office Strain Assessment (ROSA), a validated observational tool designed to assess risk factors associated with office workstation setup. The ROSA score is calculated based on chair design, monitor height, keyboard/mouse position, posture, and duration of exposure to each risk factor. Higher scores indicate greater ergonomic risk. Changes in ROSA scores will be compared between groups to determine whether the interventions improve workstation ergonomics and reduce musculoskeletal risk factors.
Lumbar Trunk Muscle Endurance Tests to measure endurance | Baseline and Week 12
  Lumbar trunk muscle endurance will be assessed using three standardized endurance tests, the unit of measurement per item will be second:
  1. Kraus-Weber Test (Trunk Flexor Endurance): Participants maintain a supported trunk flexion position while time to fatigue is recorded.
  2. Sorensen Test (Trunk Extensor Endurance): Participants maintain a horizontal torso position while the pelvis is secured, with hold time recorded.
  3. Shirado Test (Abdominal and Lumbar Endurance): Participants perform an isometric abdominal and lumbar hold, and duration until fatigue is measured.
  Longer hold times indicate better muscle endurance. Changes in endurance times will be compared between groups to determine the effectiveness of the interventions.
Surface Electromyography (sEMG) to measure muscle fatigue | Baseline and Week 12
  Muscle fatigue will be assessed using surface electromyography (sEMG) recorded from the lumbar extensor muscles during a standardized isometric contraction task. sEMG signals will be analyzed for median frequency (MF) and root mean square (RMS) changes. A decrease in MF and an increase in RMS over time indicate greater muscle fatigue. Differences in sEMG-derived fatigue indicators will be compared between intervention groups to determine the effect of the programs on lumbar muscle fatigue. The unit of measurement will be microvolts (µV).
Sit-and-Reach Test to measure flexibility | Baseline and Week 12
  Flexibility will be assessed using the Sit-and-Reach Test, which measures hamstring and lower back flexibility. Participants sit on the floor with legs extended and reach forward along a standardized measurement box. The distance reached (in centimeters) is recorded, with greater reach indicating better flexibility. Changes in Sit-and-Reach scores will be compared between groups to evaluate the effects of the interventions on flexibility. The unit of measurement will be centimeters.

CONTACTS AND LOCATIONS:
Overall Officials: Suci Wahyu Ismiyasa, M.Erg, Principal Investigator — Universiti Teknologi Mara; Zarina Zahari, PhD, Study Director — Universiti Teknologi Mara
Locations (1):
- Universitas Pembangunan Nasional Veteran Jakarta, Depok, West Java, Indonesia

IPD SHARING:
Plan to Share IPD: No